CLINICAL TRIAL: NCT05803395
Title: Incidence of Severe COVID-19 Infection in Patients With Chronic Lymphocytic Leukemia or Indolent B-cell Non-Hodgkin Lymphoma Who Received Pre-exposure Prophylaxis With Tixagevimab and Cilgavimab in Italy: an Observational Study by the GIMEMA Working Party on Chronic Lymphoproliferative Disorders and by the Fondazione Italiana Linfomi
Brief Title: Incidence of Severe COVID-19 Infection in Patients With CLL or B-NHL Who Received Pre-exposure Prophylaxis With Tixagevimab and Cilgavimab in Italy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: Fondazione Italiana Linfomi (Unknown)
Responsible Party: Sponsor
Other Study IDs: CLL2423
Record Dates: First submitted 2023-04-06; First posted 2023-04-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Lymphocytic Leukemia; Indolent B-Cell Non-Hodgkin Lymphoma; COVID-19
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational retrospective and prospective multicenter study aimed at describing the role of the COVID -19 prophylaxis with Tixagevimab and Cilgavimab in CLL or indolent B-NHL patients who received first COVID-19 prophylaxis dose between March 2022 and October 2022.

DETAILED DESCRIPTION:
This is an observational retrospective and prospective multicenter study aimed at describing the role of the COVID -19 prophylaxis with Tixagevimab and Cilgavimab in CLL or indolent B-NHL patients.

All CLL or indolent B-cell NHL patients (follicular lymphoma, marginal zone lymphoma, lymphoplasmacytic lymphoma) who received first COVID-19 prophylaxis dose with Tixagevimab and Cilgavimab according to AIFA indication between March 2022 and October 2022 will be included in the study.

Each patient will be followed for a maximum of 12 months from the first COVID-19 prophylaxis dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient with CLL or indolent B-NHL who received the first COVID-19 prophylaxis dose with Tixagevimab and Cilgavimab as per label indication between March 2022 and October 2022.
3. Signed informed consent, if applicable

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CLL or indolent B-NHL (follicular lymphoma, marginal zone lymphoma, lymphoplasmacytic lymphoma) who received the Tixagevimab and Cilgavimab as per Agenzia Italiana del Farmaco (AIFA) indications.
Sampling Method: Non-Probability Sample
Enrollment: 954 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Assess the percentage of patients who develop severe COVID-19 infection | at 12 months
  Evaluation of prophylaxis efficacy in terms of percentage of patients with CLL or indolent B-NHL who develop severe COVID-19 infection, defined as COVID-19-related hospitalization or COVID -19 related death

CONTACTS AND LOCATIONS:
Overall Officials: Gian Matteo Rigolin, Principal Investigator — Ematologia - Azienda Ospedaliero Universitaria S.Anna di Ferrara
Locations (15):
- Italy (15):
  - UOC Ematologia AO Cosenza, Cosenza
  - Ematologia AOU S.Anna, Ferrara
  - Ematologia AOU Careggi, Florence
  - ASST Lecco Ospedale A.Manzoni, Lecco
  - UOC Ematologia ATMO, Livorno
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - SCDU Ematologia, Novara
  - Dipartimento Oncologico La Maddalena, Palermo
  - UOC DI ONCOEMATOLOGIA AOR Villa Sofia - Cervello, Palermo
  - Ematologia Università "Sapienza" Roma, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - UOC Ematologia Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - SCDU Ematologia e terapie cellulari AO Mauriziano, Torino
  - Ematologia Ospedale S.Chiara, Trento
  - UOC ematologia ULSS2 Marca Trevigiana, Treviso